CLINICAL TRIAL: NCT04816058
Title: Reliability and Validity of the Turkish Version of the Ankle Instability Instrument
Brief Title: Turkish Version of the Ankle Instability Instrument
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Other Study IDs: ATADEK-2021-05/09
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankle Instability Group: Patients with a history of ankle instability or injury.
  Interventions: Behavioral: Determining the level of ankle instability
- Healthy Group: Participants without a history of ankle injury
  Interventions: Behavioral: Determining the level of ankle instability

INTERVENTIONS:
Behavioral: Determining the level of ankle instability — Ankle instability

SUMMARY:
This study aimed to translate the Ankle Instability Instrument into Turkish language, to perform a cultural adaptation study and to evaluate its validity and reliability in the Turkish population. Ankle Instability Instrument was developed to determine the ankle instability level of individuals with a history of ankle injury. Assessment of ankle instability is particularly useful in determining the complaints and functional levels of individuals with a history of functional or chronic ankle instability. It is anticipated that introducing this scale to our language will contribute to other studies in this field.

ELIGIBILITY:
Inclusion Criteria:

* History of ankle injury or sprain at least one time
* Aged between 18 to 40 years

Exclusion Criteria:

* Neurological or orthopedic disorders that may affect ankle instability.

Inclusion criteria for healthy population are; no history of ankle injury or sprain before and. aged between 18 to 40 years

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with a history of ankle injury and healthy population.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Ankle Instability Instrument | 2 weeks
  The Ankle Instability Instrument includes 9 questions that can be answered with yes or no. The first version was developed with 21 questions and later modified into 9 questions. The Ankle Instability Instrument determines the development of functional ankle instability in individuals with an ankle injury. The International Ankle Consortium reported that answering yes to 5 of 9 questions will confirm the presence of functional ankle instability. There are French and Iran versions of the Ankle Instability Instrument.
Cumberland Ankle Instability Tool | 1 day
  The ankle instability levels of the participants included in the study will be determined by the Cumberland Ankle Instability Tool. The Cumberland Ankle Instability Tool is a self-assessment scale that determines the presence of functional or chronic ankle instability and the severity of the instability. This scale consists of 9 items and the total score varies between 0 and 30. Lower scores indicate more severe instability.

SECONDARY OUTCOMES:
Short Form 12 | 1 day
  Short Form 12 is a valid and reliable scale for determining the level of quality of life. This scale consists of 12 items and can be scored as 8 subscales. These subscales are; physical function, restricted roles due to physical problems, pain, general health, energy / vitality, social functions and mental health with restricted roles due to mental problems. All items are evaluated with a 5-point Likert-type scale, and higher scores indicate better quality of life while lower scores indicate poor quality of life. This scale is used to evaluate the quality of life of healthy individuals with any pathology. Short Form 12 can be scored between 0-100 for each domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No